CLINICAL TRIAL: NCT05409469
Title: Clinical Characteristics, Management Patterns and Outcomes of Type A Aortic Dissection: A Sino-US Comparative Cohort Analysis
Status: Completed | Type: Observational
Sponsor: Xin Chen (Other)
Collaborators: China Medical University, China (Other)
Responsible Party: Sponsor-Investigator, Xin Chen, Clinical Professor, Nanjing First Hospital, Nanjing Medical University
Organization: Nanjing First Hospital, Nanjing Medical University (Other)
Other Study IDs: NanjingFirst AAD
Record Dates: First submitted 2022-05-20; First posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-05

CONDITIONS: Aortic Dissection
Keywords: Aortic Dissection; China; the United States
MeSH Terms: conditions — Aortic Dissection | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chinese patients with aortic dissection: Clinical characteristics, management patterns and outcomes of type A aortic dissection in China.
  Interventions: Procedure: surgery
- American patients with aortic dissection: Clinical characteristics, management patterns and outcomes of type A aortic dissection in the United States.
  Interventions: Procedure: surgery

INTERVENTIONS:
Procedure: surgery — surgery on patients with aortic dissection

SUMMARY:
This study constructed a retrospective cohort study by retrospectively analyzing the data of all patients with aortic dissection from January 1, 2012 to December 31, 2021 from the Cardiovascular Disease Registration System of Jiangsu Province in China and the data of similar diseases in recent years from National Inpatient Sample database in the United States

ELIGIBILITY:
Inclusion Criteria:

1.Clinical diagnosis of type A Aortic Dissection

Exclusion Criteria:

1. age<18, age unknown,
2. diagnosis of aortic aneurysm, transfer out within 1 day,
3. unknown vital status at discharge;
4. unknown treatment type: cardioplegia, valve or cardiac repair only without aortic repair or two types of treatments on different days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with aortic dissection in Jiangsu Aortic Registry system of China from January 2012 to December 2021 and all patients with aortic dissection in National Inpatient Sample database of the United States from January 2015 to December 2019.
Sampling Method: Probability Sample
Enrollment: 11550 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Baseline data of patients with type A aortic dissection was assessed by SPSS 17.0 | from 2015 to 2019
  Baseline data of patients with type A aortic dissection included gender, age,height, weight, past medical history, family history, hospital costs, etc.
The main efficacy indicators was assessed by SPSS 17.0. | from 2015 to 2019
  The main efficacy indicators included surgical procedures, surgical outcome (postoperative bleeding, ICU stay, extubation time), perioperative complications (including infection, bleeding, neurological complications, cardic complications, renal insufficiency, etc.), and postoperative mortality.

IPD SHARING:
Plan to Share IPD: No